CLINICAL TRIAL: NCT05720234
Title: The Efficacy and Safety Study of Avatrombopag Combined With IST as First-line Treatment for Severe Aplastic Anemia, A Single-arm, Phase II Clinical Study
Brief Title: Avatrombopag Combined With IST as First-line Treatment for SAA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVA&IST-001
Record Dates: First submitted 2023-01-11; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-11

CONDITIONS: Severe Aplastic Anemia
Keywords: avatrombopag
MeSH Terms: conditions — Anemia, Aplastic | interventions — avatrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): 53 subjects will be enrolled with the indicated treatment dose of avatrombopag.
  Interventions: Drug: avatrombopag

INTERVENTIONS:
Drug: avatrombopag — Patients with body weight ≥50kg were given 60mg/day and patients with body weight < 50kg were given 40mg/day for 12 weeks.
  Other Names: AVA; APAG

SUMMARY:
This single-center study aims to evaluate the early efficacy and safety of avatrombopag combined with immunosuppressive therapy (IST) in the first-line treatment of severe aplastic anemia (SAA).

DETAILED DESCRIPTION:
This is a single center, single arm, phase II clinical study. Fifty-three patients will be enrolled.

Treatment protocol is as follows: 1) Anti-human thymocyte porcine immunoglobulin (P-ATG 20mg/kg/d) or rabbit anti human thymocyte globulin (R-ATG 3.0mg/kg/d) was administered intravenously for 5 days; 2) Cyclosporine (CSA) is given at 3-5 mg/kg.d in divided doses for at least 6 months. The trough concentration is maintained at 150-250 ng/ml. 3) Avatrombopag is given orally at 60 mg once a day for patients with body weight ≥ 50 kg, and 40 mg orally once a day for patients with body weight<50 kg, for a total of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed severe aplastic anemia.
2. Men and women aged between 12 and 60.
3. Subjects must complete all screening assessments as outlined in the test protocol.
4. Able to swallow or administer orally.
5. Before the start of the research procedure, the patient or guardian should fully understand the research procedure and purpose and sign the informed consent form. If the patient's signature is not conducive to the treatment of the disease, the patient's immediate family should sign the informed consent form.

Exclusion Criteria:

1. Congenital bone marrow failure (eg. Fanconi anemia).
2. Accompanied by cytogenetic cloning changes (chromosomal karyotype and FISH detection found somatic cloning abnormalities; Simple -Y abnormality can be included in this study;) .
3. ATG or middle/high-dose cyclophosphamide was used in the past.
4. Previous treatment with cyclosporine or tacrolimus > 6 months.
5. The total course of treatment with TPO receptor agonists (including thrombopoietin, eltrombopag,hetrombopag and avatrombopag) was more than 1 month.
6. Serious infectious diseases (tuberculosis without effective control, pulmonary aspergillosis, viral infections).
7. AIDS patients.
8. Pregnant or breastfeeding, fertile but unwilling to take effective contraceptive measures.
9. Patients with malignant tumors who are not suitable for ATG treatment.
10. A newly diagnosed history of cardio/cerebral vascular thrombosis within 12 months.
11. Those who are assessed as unsuitable for inclusion by the investigator.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Treatment response | From the start of study treatment (Day1) to end of week 12.
  Percentage of patients who achieves complete response(CR) at 12 weeks.

SECONDARY OUTCOMES:
Treatment response | From the start of study treatment (Day1) to end of week 12.
  Percentage of patients achieving hematologic response (OR) at 12 weeks.
Treatment response | From the start of study treatment (Day1) to end of week 24.
  Percentage of patients achieving hematologic response and complete response (OR and CR) at 24 weeks.
Supportive treatment | From the start study treatment (Day1) up to transfusion independence.
  The time of red blood cell or platelet recovery to transfusion independence.
Incidence of Treatment-Emergent Adverse Events by CTCAE | From the start study treatment (Day1) up to week 12.
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Dose-effect relationship | From the start study treatment(Day1) up to week 24.
  Correlation between avatrombopag's serum concentration with total and complete hematological response rate.
Change of CD34+ cell | From the start study treatment(Day1) up to end of week 12 and 24.
  Change of CD34+ cells' proportion in bone marrow before and after avatrombopag treatment at week 12 and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Zhao, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No